CLINICAL TRIAL: NCT04427800
Title: An Exploration of People's Perceptions of Undergoing Treatment for Advanced Chronic Kidney Disease: a Comparison Between Different Treatment Modalities
Brief Title: Peoples Perceptions of Forms of Renal Replacement Therapy
Status: Completed | Type: Observational
Sponsor: University of Portsmouth (Other)
Collaborators: Portsmouth Hospitals NHS Trust (Other Government); University of Reading (Other)
Responsible Party: Principal Investigator, Dr Zoe Saynor, Senior Lecturer in Physical Activity, Exercise and Health, University of Portsmouth
Other Study IDs: 005JA
Record Dates: First submitted 2020-06-04; First posted 2020-06-11 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- CKD G4: Chronic kidney disease stage (G4). (eGFR < 30 mL/min/1.73m2)
- CKD G5: Chronic kidney disease stage (G5). (eGFR < 15 mL/min/1.73m2) with imminent initiation of RRT
- ESRD on ICHD: End stage renal disease on in centre haemodialysis
- ESRD on HHD: End stage renal disease on home haemodialysis
- ESRD on PD: End stage renal disease on peritoneal dialysis
- Post-transplant: Participants post-transplant

SUMMARY:
Chronic kidney disease (CKD) causes symptoms and potential loss of independence. These effects are increased as the disease progress to endstage renal disease (ESRD), particularly when external intervention (i.e.

dialysis) is used to keep these individuals alive. The combined effect of ESRD and its treatment has a significant impact on an individual's life, potentially causing reduced employment time, reduced social time and increased anxiety/stress.

The purpose of this study is to investigate the impact that CKD/ESRD have on an individual's life. Specifically, this study is focused on giving an insight into the psychosocial impact that CKD/ESRD and different forms of renal replacement therapy have upon these individuals.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) affects over 4% of the UK population, with approximately 118 per million population commencing treatment for end-stage kidney disease each year (UK renal registry, 2017). As enal function deteriorates, these individuals become progressively symptomatic and require renal replacement therapy (RRT). CKD is split into five stages, classified by their glomerular filtration rate (eGFR), with stages G4 and G5 representing advanced disease preceding end-stage renal failure (Levey et al., 2005).

Along with diminished physical ability, cognitive function and quality of life (QoL) have also been shown to deteriorate within this population (Abdel-Kader, Unruh, & Weisbord, 2009).

Previous findings have shown that individuals with renal disease, particularly advanced CKD/ESRD have a reduced QoL and substantial symptom burden, defined as a loss of functional abilities along with psychological suffering affected by the impact of their symptoms (Gill, Chakraborty, & Selby, 2012). Of note, this seems to become particularly notable at the initiation of RRT (Pagels, Söderkvist, Medin, Hylander, & Heiwe, 2012). This supports previous findings by Davison & Jhangri (2010) and findings by Lowney et al (2015) who found that individuals undergoing in-centre haemodialysis (HD) had a substantial symptom burden which was associated with a reduced health-related QoL. This is significant because in-centre HD (ICHD) is currently the most common form of RRT globally.

To date, no research has qualitatively examined the burden of other forms of RRT, such as home haemodialysis (HHD), which is typically undertaken at home more frequently and for shorter durations than ICHD; and peritoneal dialysis (PD), where the peritoneum is used as a membrane through which excess fluid and toxins are removed from the body. A recent investigation by Jones and colleagues (2018) explored the perceptions of UK-based individuals undergoing ICHD within the National Health Service (NHS). Interestingly, several common themes were identified; including fluctuations in their QoL and well-being over the course of their HD therapy and restrictions in their social lives, due to HD scheduling and the heavy emotional impact on themselves and others. These were shown to often be overlooked in the literature, however, these factors have the potential to negatively impact an individual's QoL and sense of self, defined as one's sense of purpose in life. Importantly, higher rates of depression and anxiety have also been reported in individuals with CKD (Chen et al., 2010; Semaan, Noureddine, & Farhood, 2018). For example, Barros et al. (2016) found that greater than 30% of individuals had depressive symptoms and reduced QoL. Furthermore, those found with depressive symptoms tended to have a lower survival rate at the 2-year evaluation period. It has been postulated that this increased prevalence in depressive symptoms could be due to some significant psychosocial implications of CKD such as, reductions in employment, social and personal time and interpersonal relationships (Finnegan-John & Thomas, 2013), supported by a recent (currently unpublished) investigation conducted by the research team for this study at the Wessex Kidney Centre (WKC). During this study, it became clear through informal discussions with people with ESRD and the treatment of this impacts their lives greatly and that qualitative markers of QoL had the potential to be very insightful into the impact of ESRD. Given the above, this study aims to investigate the QoL of adults at the advanced stages of CKD (CKD stage G4 and G5) and those on all modalities of RRT (ICHD, HHD, PD, and transplantation).

ELIGIBILITY:
Inclusion Criteria:

Aged 18 years or older Willing and able to undertake the interview process Able to give informed consent

Exclusion Criteria:

Age < 18 years Does not provide written informed consent Any neurological/psychiatric diagnoses Lack of fluency in English Individuals who have commenced RRT within three months of the study start date Transplant patients being seen in clinic more than once every fortnight

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults with advanced CKD/ESRD (eGFR < 30 mL/min/1.73m2
  ) will be recruited into this study. Persons falling into six distinct categories will be approached:
  1. CKD G4
  2. CKD G5 with imminent initiation of RRT
  3. ESRD on ICHD
  4. ESRD on HHD
  5. ESRD on PD
  6. Post-transplant
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2020-11-24 (Actual)

PRIMARY OUTCOMES:
Thematic analysis of qualitative interview exploring the experiences of renal disease and renal replacement therapy in adults with advanced chronic kidney disease and end-stage renal disease | Day 1
  Qualitative interviews to explore the above experiences

CONTACTS AND LOCATIONS:
Locations (1):
- School of Sport Health and Exercise Science, Portsmouth, Outside the United States Or Canada, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Transcripts will not be uploaded to a repository